CLINICAL TRIAL: NCT01505296
Title: Randomized Comparison of Catheter Ablation Versus Anti-arrhythmic Drug Therapy in Patients With Recently Diagnosed Paroxysmal Atrial Fibrillation as Assessed by a Continuous Implantable Monitor
Brief Title: Catheter Ablation for Recently Diagnosed Paroxysmal Atrial Fibrillation
Acronym: CABAL
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Never initiated
Sponsor: Valley Health System (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Jonathan Steinberg,MD, Director Arrhythmia Services, Valley Health System, Valley Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BWI-IIS-0143
Record Dates: First submitted 2011-12-28; First posted 2012-01-06 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Atrial Fibrillation
Keywords: Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anti-Arrhythmia Agents; Flecainide; Sotalol; dofetilide; Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antiarrhythmic drug (Active Comparator): Class I or III antiarrhythmic drug
  Interventions: Drug: Antiarrhythmic drug
- Catheter ablation (Experimental): Pulmonary vein isolation
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Drug: Antiarrhythmic drug — propafenone, flecainide, sotalol, dofetilide
  Other Names: Rhythmol, Tambocor, Betapace, Tikosyn
  Arms: Antiarrhythmic drug
Procedure: Catheter ablation — Complete PVI
  Other Names: Thermocool
  Arms: Catheter ablation

SUMMARY:
The objective is to compare the progression of Atrial Fib (AF) burden by continuous monitoring in patients with recently diagnosed paroxysmal AF treated by catheter ablation (PVI) versus anti-arrhythmic drug (AAD) therapy.

DETAILED DESCRIPTION:
Randomized, multicenter clinical trial comparing medical therapy (Group I) with ablation therapy(Group II). Randomization will be determined by opening a sealed envelope. All patients will be implanted with an implantable loop recorder and followed every three months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recently diagnosed paroxysmal AF who are eligible to receive specific rhythm control therapy

Exclusion Criteria:

* Previous treatment with Class IC or class III AAD
* Previous AF ablation procedure
* Congestive heart failure (NYHA III-IV functional class)
* Left Ventricle ejection fraction less than 35%
* Left atrial diameter > 55mm
* Unwillingness to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percentage of AF burden | 4 months
  The percentage of AF burden defined through continuous monitoring using an implnatage loop recorder (ILR)

SECONDARY OUTCOMES:
All-death death | 4 months
  All-cause death, thromboembolic events, hospitalizations, procedural complications, drug adverse effects, and number of crossovers

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Steinberg, MD, Principal Investigator — Valley Health System; Evegny Pokushalou, MD, Principal Investigator — State Resarch Institute of Circulation Pathology, Novosibirsk, Siberia
Locations (2):
- Valley Health System, Ridgewood, New Jersey, United States
- State Research Institute of Circulation Pathology, Novosibirsk, Russia